CLINICAL TRIAL: NCT04094298
Title: Use of Extended Release Triamcinolone in the Treatment of Rotator Cuff Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0258
Record Dates: First submitted 2019-08-07; First posted 2019-09-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Tendinitis; Rotator Cuff Impingement; Injections; Glucocorticoids
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome | interventions — FX006

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Patients receiving the 32-unit injection of FX006.
  Interventions: Drug: FX006 Injection

INTERVENTIONS:
Drug: FX006 Injection — One injection of extended release triamcinolone. 32 milligram injection of the extended release triamcinolone in a 75:25 ratio of polylactic-co-glycolic acid (PLGA) microspheres to drug load of 25%. The drug product is reconstituted with diluent containing an isotonic, sterile aqueous solution of sodium chloride, carboxymethylcellulose sodium and polysorbate-80 to form a suspension prior to injection.
  Other Names: No other interventions

SUMMARY:
The primary objective of this study is to assess the overall safety and general tolerability of extended release triamcinolone acetate (TA-ER/FX006) in patient with rotator cuff disease. The study will enroll 65 patients, aged 40-75 years old, in a longitudinal case series level IV study using extended release triamcinolone to treat shoulder pain from rotator cuff disease. Inclusion criteria will be shoulder pain without a history of trauma and physical exam consistent with rotator cuff tendinitis, impingement syndrome or rotator cuff tear.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and efficacy of TA-ER in the treatment of rotator cuff disease. The study will enroll 65 patients in a longitudinal case series level IV study using extended release triamcinolone to treat shoulder pain from rotator cuff disease. Inclusion criteria will be shoulder pain without a history of trauma and physical exam consistent with rotator cuff tendinitis, impingement syndrome or rotator cuff tear. Patients will have normal Xrays or Xrays indicative of chronic cuff tearing and a musculoskeletal ultrasound indicating an intact rotator cuff, partial cuff tearing or cuff tear. Patients will undergo an ultrasound guided injection of TA-ER into the subacromial space from a lateral access point at the time of the examination. They will be monitored for any immediate adverse effects. Patient reported outcomes measures will be recorded with online questionnaires which include a Visual Analog Scale (VAS), Single assessment numeric evaluation (SANE), Veteran's Rand 12 (VR-12) and American Shoulder and Elbow Scale (ASES) and will be recorder pre-treatment and at 2, 4, 8 and 12 and 24 weeks post treatment. Patients will be asked to follow up for an in person evaluation at 4 weeks, 12 weeks and 24 weeks post injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 40-75 years old.
2. Able and willing to give written informed consent in accordance with the IRB.
3. Read and Speak English.
4. History indicative of rotator cuff disease.
5. Physical exam consistent with rotator cuff disease.
6. All patients will have AP and Outlet X ray views.
7. X rays will be normal or indicative of chronic RTC tearing
8. Musculoskeletal Ultrasound indicating intact RTC, full thickness tears, or large and massive cuff tears in older, sedentary individuals.
9. Willing to abstain from use of NSAIDs

Exclusion Criteria:

1. Females who are pregnant or nursing or plan to become pregnant during the study; men who plan to conceive during the study; or unwilling to practice birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Known or suspected hypersensitivity to FX006 (or component of FX006), triamcinolone acetonide.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 24 weeks
  Assess the overall safety extended release triamcinolone in acetate (TA-ER/FX006) in patient with rotator cuff disease. Safety is evaluated on the basis of incidence of adverse events (AE). These would be reported by the patient or discovered by the investigator from the following measure below: VAS (Visual Analogue Scale) is a scale to measure patient's pain. SANE (Single Assessment Numeric Evaluation) a scale of 0 to 100 that patients rate their joint function, with 100 being normal function. VR12 (Veterans RAND 12 Item Health Survey) is a patient-reported measure of a patient's overall health. ASES (American Shoulder and Elbow Surgeons Standardized Shoulder Assessment) is a survey which measures function and pain in the shoulder. Surveys could indicate an AE if there was increasing pain or worsening function which would not be expected. This would direct the investigator into further physical exam and inquiry on possible injuries or any other AE. Outcomes will not be aggregated.

SECONDARY OUTCOMES:
Change in shoulder pain as assessed by VAS | 24 weeks
  Assess changes in shoulder pain. Change in shoulder pain as measured by VAS. The VAS (Visual Analogue Scale for pain) is a continuous scale to measure patient's pain. The scale is from 0 to 100 with 100 being the worst pain and 0 being no pain.
Change in shoulder function as assessed by SANE | 24 weeks
  Assess changes in shoulder function. Change in shoulder function as measured by SANE. SANE (Single Assessment Numeric Evaluation) is a scale of 0 to 100 that patients rate their knee function, with 100 being normal function and 0 being no function.
Change in shoulder function as assessed by VR-12 | 24 weeks
  health. It includes 12 questions which correspond to seven health domains: general health, physical function, limitations due to physical and emotional problems, bodily pain, energy level, social functioning, and mental health. There are two scores from the VR-12, a Mental Component Score and a Physical Component Score. The scores are reported as Z-scores (number of standard deviations away from population average). The average score for the United States population is 50 and 1 standard deviation corresponds to 10 points.
Change in shoulder function and pain as assessed by ASES | 24 weeks
  ASES (American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form) is a patient reported questionnaire which measures function and pain in the shoulder. This is a 100 point scale that combines 50 points from pain and 50 points from function. There are 2 sections to the form: pain and activities of daily living. The pain section has 4 yes or no questions regarding timing of pain and pain medication, and 1 question involving a VAS scale from 0 (no pain) to 10 (worst pain). The activities of daily living section has 10 questions and is ranked on a 0 (unable to perform) to 3 (no difficulty performing) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Camhi, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Orthopedic Institute at Great Neck, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conaghan PG, Hunter DJ, Cohen SB, Kraus VB, Berenbaum F, Lieberman JR, Jones DG, Spitzer AI, Jevsevar DS, Katz NP, Burgess DJ, Lufkin J, Johnson JR, Bodick N; FX006-2014-008 Participating Investigators. Effects of a Single Intra-Articular Injection of a Microsphere Formulation of Triamcinolone Acetonide on Knee Osteoarthritis Pain: A Double-Blinded, Randomized, Placebo-Controlled, Multinational Study. J Bone Joint Surg Am. 2018 Apr 18;100(8):666-677. doi: 10.2106/JBJS.17.00154. PMID 29664853
- [Background] Gaujoux-Viala C, Dougados M, Gossec L. Efficacy and safety of steroid injections for shoulder and elbow tendonitis: a meta-analysis of randomised controlled trials. Ann Rheum Dis. 2009 Dec;68(12):1843-9. doi: 10.1136/ard.2008.099572. Epub 2008 Dec 3. PMID 19054817
- [Background] Tashjian RZ, Deloach J, Green A, Porucznik CA, Powell AP. Minimal clinically important differences in ASES and simple shoulder test scores after nonoperative treatment of rotator cuff disease. J Bone Joint Surg Am. 2010 Feb;92(2):296-303. doi: 10.2106/JBJS.H.01296. PMID 20124055
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Result] Jain NB. Do These Crystals Really Sparkle?: Commentary on an article by Philip G. Conaghan, MBBS, PhD, FRACP, FRCP, et al.: "Effects of a Single Intra-Articular Injection of a Microsphere Formulation of Triamcinolone Acetonide on Knee Osteoarthritis Pain. A Double-Blinded, Randomized, Placebo-Controlled, Multinational Study". J Bone Joint Surg Am. 2018 Apr 18;100(8):e56. doi: 10.2106/JBJS.17.01520. No abstract available. PMID 29664865